CLINICAL TRIAL: NCT01921855
Title: A Phase I, Randomized, Double-blind, Placebo Controlled, Single Dose Escalation Study of FVIIa Variant BAY86-6150 (B0189) in Subjects With Moderate or Severe Hemophilia Types A or B With or Without Inhibitors
Brief Title: Study of FVIIa Variant BAY86-6150 (B0189) in Subjects With Moderate or Severe Hemophilia Types A or B With or Without Inhibitors
Acronym: MATCHBOX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 13787; 2008-000117-29 (EudraCT Number)
Record Dates: First submitted 2013-07-10; First posted 2013-08-13 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Hemophilia A; Hemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- BAY Factor VII (6.5 µg/kg) / Placebo (Experimental): n = 4, randomized 3:1; 6.5 µg/kg BAY 86-6150 (B0189):Placebo
  Interventions: Drug: BAY Factor VII (BAY86-6150); Drug: Placebo
- BAY Factor VII (20 µg/kg) / Placebo (Experimental): n = 4, randomized 3:1; 20 µg/kg BAY 86-6150 (B0189):Placebo
  Interventions: Drug: BAY Factor VII (BAY86-6150); Drug: Placebo
- BAY Factor VII (50 µg/kg) / Placebo (Experimental): n = 4, randomized 3:1; 50 µg/kg BAY 86-6150 (B0189):Placebo
  Interventions: Drug: BAY Factor VII (BAY86-6150); Drug: Placebo
- BAY Factor VII (90 µg/kg) / Placebo (Experimental): n = 4, randomized 3:1; 90 µg/kg BAY 86-6150 (B0189):Placebo
  Interventions: Drug: BAY Factor VII (BAY86-6150); Drug: Placebo

INTERVENTIONS:
Drug: BAY Factor VII (BAY86-6150) — BAY Factor VII (BAY86-6150), 6.5 µg/kg body weight, will be administered as a slow intravenous (i.v.) administration over a period of 2-5 minutes (min) on Study Day 1.
  Arms: BAY Factor VII (6.5 µg/kg) / Placebo
Drug: BAY Factor VII (BAY86-6150) — BAY Factor VII (BAY86-6150), 20 µg/kg body weight, will be administered as a slow intravenous (i.v.) administration over a period of 2-5 minutes (min) on Study Day 1.
  Arms: BAY Factor VII (20 µg/kg) / Placebo
Drug: BAY Factor VII (BAY86-6150) — BAY Factor VII (BAY86-6150), 50 µg/kg body weight, will be administered as a slow intravenous (i.v.) administration over a period of 2-5 minutes (min) on Study Day 1.
  Arms: BAY Factor VII (50 µg/kg) / Placebo
Drug: BAY Factor VII (BAY86-6150) — BAY Factor VII (BAY86-6150), 90 µg/kg body weight, will be administered as a slow intravenous (i.v.) administration over a period of 2-5 minutes (min) on Study Day 1.
  Arms: BAY Factor VII (90 µg/kg) / Placebo
Drug: Placebo — Placebo will be administered as a slow intravenous (i.v.) administration over a period of 2-5 minutes (min) on Study Day 1.

SUMMARY:
This is the first in humans study of BAY86-6150 (B0189) in non-bleeding subjects with moderate or severe congenital hemophilia A or B with or without inhibitors. This is a randomized, double-blind, placebo-controlled, single-dose, dose escalation study. It is designed to investigate the safety, tolerability, potential immunogenicity, pharmacokinetic and pharmacodynamic profile of BAY86-6150 (B0189) and to determine a dose or range of doses to be examined in subsequent studies.

ELIGIBILITY:
Inclusion Criteria:

* History of moderate or severe congenital hemophilia A or B with or without inhibitors to Factor VIII (FVIII) or Factor IX (FIX)
* Male subjects 18-65 years of age inclusive
* Able to dismiss factor replacement therapy during the course of the study unless required for the treatment of an acute bleeding episode
* Written informed consent
* Willing and able to comply with the requirements of the protocol
* Have adequate venous access
* Willing to use an effective method of contraception until Day 30 of their study participation

Exclusion Criteria:

* Received factor replacement therapy or treatment with any other procoagulant therapeutics, or any antifibrinolytic agents, including blood products, at anytime within 5 days prior to administration of investigational medicinal product (IMP)
* Planned administration of factor replacement therapy or treatment with any other procoagulant therapeutics or any antifibrinolytic agents, including blood products, at anytime during the study period
* Acute bleeding episode or any ongoing bleeding episode at any time within 7 days prior to administration IMP
* Clinically relevant coagulation disorder other than congenital hemophilia A or B
* History of angina or receiving treatment for angina
* History of coronary atherosclerotic disease, disseminated intravascular coagulopathy, or stage 2 hypertension defined as systolic blood pressure (SBP) >/= 160 mmHg or diastolic blood pressure (DBP) >/= 90 mmHg
* History of transient ischemic attack, stroke, myocardial infarction, coronary artery disease, congestive heart failure, or thromboembolic event
* Active infection on day of IMP administration or septicemia at any time within 30 days prior to administration of IMP

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Up to Day 50

SECONDARY OUTCOMES:
Pharmacokinetic assessment, based on plasma concentration of BAY86-6150 | 9 time points from pre-dosing on Day 1 up to 48 hours post-dosing
Pharmacodynamic assessment, based on plasma hemostasis marker level | 9 time points from pre-dosing on Day 1 up to 48 hours post-dosing
Immunogenicity assessment, based on anti-BAY86-6150 binding antibody levels | 3 time points from pre-dosing on Day 1 up to Day 50

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- Warsaw, Poland
- South Africa (2):
  - Bloemfontein, Freestate
  - Johannesburg, Gauteng
- London, United Kingdom

REFERENCES:
- [Result] Mahlangu JN, Coetzee MJ, Laffan M, Windyga J, Yee TT, Schroeder J, Haaning J, Siegel JE, Lemm G. Phase I, randomized, double-blind, placebo-controlled, single-dose escalation study of the recombinant factor VIIa variant BAY 86-6150 in hemophilia. J Thromb Haemost. 2012 May;10(5):773-80. doi: 10.1111/j.1538-7836.2012.04667.x. PMID 22353395